CLINICAL TRIAL: NCT00382330
Title: Chemoprevention of Cancer in the Lower Female Genital Tract: The Antineoplastic Activity of the Fungicide Ciclopirox.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0120050348
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-04

CONDITIONS: Vulvar Cancer
Keywords: Vulva
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Ciclopirox

INTERVENTIONS:
Drug: Ciclopirox

SUMMARY:
The purpose of this study is to determine if regular and daily repeated application of the ciclopirox lotion to vulva will make the precancerous lesion(s) shrink or even disappear.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages 18 and 75 years.
* Patients may be carriers of the Human Immunodeficiency Virus (HIV).
* Patients must have been diagnosed with precancerous lesion(s) of the vulva by tissue sampling (biopsy-proven vulvar intraepithelial neoplasia grade II or III)
* Patients must be able to come to University Hospital for their initial appointment in Gynecologic Oncology Clinic, and for the eight follow-up visits in that Clinic required by the protocol.

Exclusion Criteria:

* Pregnant or patients who are breast feeding a baby.
* Patients who have been diagnosed with a vaginal yeast infection.
* Patients who have undergone prior surgery for precancerous lesion(s) of the vulva.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Cracchiolo, MD, MPH, Principal Investigator — University of Medicine and Dentistry of New Jersey
Locations (1):
- University of Medicine and Dentistry of NJ, Newark, New Jersey, United States